CLINICAL TRIAL: NCT07272317
Title: PSMA-PET/MRI-Ultrasound Multimodal Fusion Navigation for Da Vinci Robot-Assisted Radical Prostatectomy: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Liu Cheng, Chief Physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 【2025】177; Y2025082 (Other Grant/Funding Number: Shanghai General Hospital Leadership Talent Program)
Record Dates: First submitted 2025-11-17; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a single-center, prospective randomized controlled trial. The research subjects are patients with T3a or T2 (with the lesion close to the surface of the prostate) prostate cancer who underwent robot-assisted radical prostatectomy (RARP) in our hospital. The subjects were randomly divided into a control group and an experimental group. Patients in the control group received RARP according to the conventional method, while patients in the experimental group underwent preoperative PSMA-PET/MRI-ultrasound multimodal fusion and RARP under real-time navigation assistance during the operation.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group（navigation-assisted RARP） (Experimental): The experimental group will use preoperative PSMA-PET/MRI and intraoperative ultrasound for multimodal fusion to construct a three-dimensional model and synchronize it in real time to the surgeon's control console through the Da Vinci surgical robot's Tilepro video integration module, and complete the anterior approach laparoscopic radical prostatectomy under this guidance.
  Interventions: Procedure: experimental group (navigation-assisted RARP)
- Control group (traditional RARP) (No Intervention): The control group will undergo the anterior approach laparoscopic radical prostatectomy in the conventional manner.

INTERVENTIONS:
Procedure: experimental group (navigation-assisted RARP) — Before the surgery, the prostate and lesions were delineated on PET/MRI: at least two nuclear medicine physicians independently reviewed the images and provided a unified report. The experimental group had the external contour of the prostate and the three-dimensional lesion schematic diagram delineated by the urologist. A BK5000 ultrasound probe was inserted into the rectum, the probe was fixed to the surgical bed frame by the stepper, and the real-time images of the prostate were captured by the ultrasound.The multimodal fusion of the three-dimensional lesion outlined by ultrasound and PSMA-PET/MRI was achieved through the built-in MIM software. Subsequently, picture-in-picture guidance was realized through the Da Vinci Tilepro functional module, and the edge of the lesion was marked with titanium clips. After the ultrasound probe was withdrawn, the peripheral resection of the prostate, nerve preserve or not were completed under the guidance of the titanium clips.
  Arms: experimental group（navigation-assisted RARP）

SUMMARY:
Radical prostatectomy faces the core dilemma of balancing functional preservation with tumor eradication. While nerve-sparing techniques improve urinary control, intraoperative tumor localization remains imprecise, resulting in positive surgical margin (PSM) rates of 11%-38% and elevated recurrence risk. Traditional preoperative 2D imaging fails to dynamically guide surgical boundaries. Although multimodal fusion studies (e.g., MRI or PSMA-PET/CT) attempt to address this, they struggle to achieve simultaneous precision in lesion identification and real-time spatial tracking. This study pioneers a PSMA-PET/MRI-ultrasound multimodal fusion navigation system for the Da Vinci surgical robot, leveraging three innovations: PSMA-PET/MRI dual-modality synergy for subclinical lesion detection at millimeter resolution; Non-rigid point-cloud registration algorithms to dynamically compensate for intraoperative prostate deformation, enabling 3D ultrasound-PET/MRI elastic fusion; Utilizing the telipro port of the Da Vinci surgical robot to achieve intraoperative picture-in-picture navigation, real-time localization of the tumor boundary, and precise resection as well as precise protection.This study aims to verify the safety and effectiveness of the world's first PSMA-PET/MRI-ultrasound multimodal fusion navigation system adapted for the Da Vinci surgical robot. This system is expected to reduce the positive margin rate to less than 10%, increase the rate of nerve preservation by 30%, shorten the postoperative urinary control recovery time to within 2 weeks, and establish a standard process for robotic surgery navigation. This will provide a new paradigm for precise surgical treatment of prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer, the second most prevalent malignancy in men globally, has long grappled with a core dilemma in radical surgery: balancing functional preservation against oncological efficacy. Although nerve-sparing techniques significantly improve postoperative urinary control and sexual function (with robotic surgery achieving >80% continence recovery rates), conventional approaches relying on intraoperative visual tumor boundary assessment result in positive surgical margin (PSM) rates of 11%- 38%, increasing biochemical recurrence risk exceeding 40% [1,2]. For locally advanced cases, sacrificing functional structures to ensure oncological radicality leads to postoperative erectile dysfunction rates up to 95% and urinary incontinence exceeding 50% [3].The essence of this conflict lies in: Extended resection reduces PSM rates but damages neurovascular bundles (NVBs) governing micturition and erectile function; Limited resection preserves function yet increases PSM risk due to residual microlesions-particularly in anatomically complex zones like the prostatic apex and anterior wall, where visual localization errors typically exceed 3 mm.

Preoperative imaging limitations exacerbate this: MRI offers high anatomical resolution (0.5 mm³) but cannot track intraoperative organ deformation; PSMA-PET/CT detects micrometastases with 98% sensitivity, yet spatial registration errors between metabolic/anatomical data exceed 2 mm [4]. Current multimodal fusion approaches are inadequate: MRI-based fusion misses early-stage lesions due to limited tumor contrast; PSMA-PET/CT fusion suffers from metabolic-anatomical misalignment.

Thus, a navigation system enabling simultaneous subclinical lesion detection and dynamic deformation compensation is imperative to resolve the function-versus-curability dilemma.

We have adopted the following approaches to complete the construction of the intraoperative navigation system: (1) On the PET/MRI before the operation, the prostate and the lesion were delineated: at least two nuclear medicine physicians independently reviewed the images and then provided a unified report; the external contour of the prostate and the three-dimensional lesion schematic diagram of the lesion were then delineated by a urologist; (2) On the intraoperative ultrasound, the prostate was delineated: the prostate image was captured in real time by BK ultrasound and then the external contour of the prostate was delineated by a urologist; (3) The multimodal fusion of the three-dimensional lesion delineated by BK ultrasound and PSMAPET/MRI was achieved through the MIM software built into the BK ultrasound; (4) The intraoperative resection was guided by the Da Vinci Tilepro functional module. So far, 6 cases have been successfully completed and compared with 6 T3a patients randomly selected from previous conventional surgeries. Currently, due to the small sample size, although the differences in the surgical margins have not reached a statistically significant difference, a trend of difference has been demonstrated. Due to the short follow-up period, the postoperative PSA and urination conditionshave not been included in the statistical cohort.

ELIGIBILITY:
Inclusion Criteria:

* Target Population: Patients with clinical stage T3a, or T2 (with the lesion close to the surface of the prostate) scheduled for robot-assisted radical prostatectomy (RARP), who have been diagnosed with prostate cancer.

  * Age 50 - 80 years old;

    * Pathologically confirmed as prostate adenocarcinoma (Gleason score 6 - 10);

      * PSMA-PET/MRI indicates extracapsular invasion of the lesion; ④ Signed informed consent and committed to completing follow-up.

Exclusion Criteria:

* ① Metastasis (M1 stage) or lymph node metastasis (N1 stage);

  * Previous pelvic radiotherapy or endocrine therapy history;

    * Severe cardiopulmonary dysfunction (ASA grade ≥ III); ④ Mental illness or cognitive impairment that cannot cooperate with assessment; ⑤ Participating in other interventional clinical trials.

Max Age: 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Positive margin rate | After being enrolled, the patient undergoes radical prostatectomy for prostate cancer. Around 7 to 10 days after the surgery, the pathological report will be available.
  Positive margin rate (prostate radical specimens need to be stained with standard ink, and the contact between tumor cells and the ink surface of the surgical specimen is considered a positive margin; two pathologists with qualifications of associate chief physician or above (who need to have 5 years of prostate pathology diagnosis experience) blind to the patient information and independently read the films， if the two interpretations are inconsistent，the third senior pathologist (senior professional title) will review) .

SECONDARY OUTCOMES:
Nerve Preservation Success Rate, as assessed by International Index of Erectile Function-5 (IIEF-5) score and maximum urine flow rate (Qmax) | Follow-up was conducted for 6 months after the surgery.
  The proportion of patients achieving nerve preservation success, defined as simultaneouslyhaving an International Index of Erectile Function-5 (IIEF-5) score ≥ 21 and a maximum urine flow rate (Qmax) ≥ 15 ml/s at 6 months after surgery
Time to Urinary Continence Recovery | Follow-up was conducted for 6 months after the surgery.
  The number of consecutive days from the date of surgery until the patient uses no more than one safety pad per day.
Serum Prostate-Specific Antigen (PSA) Level | Follow-up was conducted for 6 months after the surgery.
  Extract the peripheral blood of patients, measure and record the PSA level (ng/ml) at 6 weeks, 3 months, and 6 months after surgery.
Biochemical Recurrence Rate as assessed by PSA level after the surgery | Follow-up was conducted for 6 months after the surgery.
  The proportion of patients with biochemical recurrence after surgery, defined as a rising PSA level (e.g., PSA ≥ 0.2 ng/mL) confirmed by a second consecutive test.
Number of participants with postoperative complications as assessed by the Clavien-Dindo classification system | Follow-up was conducted for 6 months after the surgery.]
  Number of participants with postoperative complications according to the Clavien-Dindo classification system.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sivarajan G, Prabhu V, Taksler GB, Laze J, Lepor H. Ten-year outcomes of sexual function after radical prostatectomy: results of a prospective longitudinal study. Eur Urol. 2014 Jan;65(1):58-65. doi: 10.1016/j.eururo.2013.08.019. Epub 2013 Aug 26. PMID 24007711
- [Background] Bakht MK, Beltran H. Biological determinants of PSMA expression, regulation and heterogeneity in prostate cancer. Nat Rev Urol. 2025 Jan;22(1):26-45. doi: 10.1038/s41585-024-00900-z. Epub 2024 Jul 8. PMID 38977769
- [Background] Zhang L, Wu B, Zha Z, Zhao H, Jiang Y, Yuan J. Positive surgical margin is associated with biochemical recurrence risk following radical prostatectomy: a meta-analysis from high-quality retrospective cohort studies. World J Surg Oncol. 2018 Jul 3;16(1):124. doi: 10.1186/s12957-018-1433-3. PMID 29970100
- [Background] Tewari A, Sooriakumaran P, Bloch DA, Seshadri-Kreaden U, Hebert AE, Wiklund P. Positive surgical margin and perioperative complication rates of primary surgical treatments for prostate cancer: a systematic review and meta-analysis comparing retropubic, laparoscopic, and robotic prostatectomy. Eur Urol. 2012 Jul;62(1):1-15. doi: 10.1016/j.eururo.2012.02.029. Epub 2012 Feb 24. PMID 22405509